CLINICAL TRIAL: NCT03544229
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Phase 2b Study to Evaluate the Efficacy and Safety of Twice-Daily Oral Administration of a Peripherally Acting Dopamine Receptor D2/D3 Antagonist, TAK-906 for the Treatment of Adult Subjects With Symptomatic Idiopathic or Diabetic Gastroparesis
Brief Title: A Study to Evaluate the Efficacy and Safety of TAK-906 in Adult Participants With Symptomatic Idiopathic or Diabetic Gastroparesis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAK-906-2002; 2018-001275-21 (EudraCT Number); U1111-1211-2779 (Other: Universal Trial Number)
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Results first posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-10

CONDITIONS: Diabetic Gastroparesis; Idiopathic Gastroparesis
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): TAK-906 maleate placebo-matching capsules, orally, twice daily (BID) for up to 12 weeks.
  Interventions: Drug: Placebo
- TAK-906 Maleate 5 mg (Experimental): TAK-906 maleate 5 mg, capsules, orally, BID for up to 12 weeks.
  Interventions: Drug: TAK-906 Maleate
- TAK-906 Maleate 25 mg (Experimental): TAK-906 maleate 25 mg, capsules, orally, BID for up to 12 weeks.
  Interventions: Drug: TAK-906 Maleate
- TAK-906 Maleate 50 mg (Experimental): TAK-906 maleate 50 mg, capsules, orally, BID for up to 12 weeks.
  Interventions: Drug: TAK-906 Maleate

INTERVENTIONS:
Drug: TAK-906 Maleate — TAK-906 maleate capsules.
  Arms: TAK-906 Maleate 25 mg; TAK-906 Maleate 5 mg; TAK-906 Maleate 50 mg
Drug: Placebo — TAK-906 maleate placebo-matching capsules.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the efficacy and safety of treatment with 2 dose levels of TAK-906 in adult participants with gastroparesis compared with placebo during 12 weeks of treatment.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-906. TAK-906 is being tested to treat people who have symptomatic idiopathic or diabetic gastroparesis.

The study will enroll approximately 205 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the three treatment groups (in 1:1:1:1 ratio) which will remain undisclosed to the patient and study doctor during the study (unless there is an urgent medical need):

* TAK-906 Maleate 5 mg (After implementation of Amendment 8, participants will not be further randomized to this arm)
* TAK-906 Maleate 25 mg
* TAK-906 Maleate 50 mg Placebo (dummy inactive pill) - this is a capsule that looks like the study drug but has no active ingredient

Prior to Amendment 8, participants were randomized to receive TAK-906 5 mg. After implementation of Amendment 8, participants will not be further randomized to this dose arm. All participants will be asked to take one capsule twice daily, at approximately the same time each day throughout the study.

This multi-center trial will be conducted worldwide. The overall study duration is approximately 17 weeks. Participants will make multiple visits to the clinic, and will be contacted by telephone 30 days after receiving their last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Should have experienced symptoms of gastroparesis (e.g., postprandial fullness, nausea, vomiting, upper abdominal pain, and early satiety for at least 3 months before screening as assessed by a physician.
2. Must have confirmed delayed gastric emptying by meeting 1 of the following criteria:

   1. Confirmed by an accepted diagnostic testing method (Gastric Emptying Breath Test [GEBT], scintigraphy, or wireless motility capsule) that is documented in the participant's medical records prior to screening; OR
   2. Participants without previous confirmation of delayed gastric emptying prior to screening will undergo a GEBT after they have stopped taking prohibited medications.
3. Must have an average composite ANMS GCSI-DD symptom score ≥2 during the 7 days before randomization. The predominant symptom experienced by participants must not be abdominal pain.
4. Must experience nausea: nausea subscale (of ANMS GCSI-DD) symptom score ≥2 at least 4 of 7 days or an average nausea subscale symptom score ≥2 during the 7 days before randomization. Nausea symptoms must not be attributable to a central disorder (e.g. motion sickness, glaucoma, menstrual cycles, migraine headache).
5. Has a body mass index (BMI) of ≥18 to ≤40 kg/m^2 inclusive.
6. Participant with diabetes mellitus must have glycosylated hemoglobin (HbA1c) ≤11% at screening and before randomization.
7. Absence of gastric outlet obstruction confirmed by upper GI, computed tomography or endoscopy.

Exclusion Criteria:

1. Known secondary causes of gastroparesis including but not limited to Parkinson disease, cancer, viral illness, or connective tissue diseases.
2. Predominant gastroparetic symptom is epigastric pain, diffuse abdominal pain, or pain associated with bowel movement.
3. Is taking medications that affect gastric emptying including opioids, glucagon-like peptide-1 analogs (e.g., exenatide, liraglutide), amylin analogs (e.g., pramlintide), and cannabinoids.
4. Prior history of gastric surgery, including but not limited to gastrectomy, gastric bypass, gastric banding, bariatric surgery, pyloroplasty, vagotomy, or fundoplication, which has manipulated the natural anatomy of the stomach.
5. History of intra-pyloric botulinum toxin injection within 3 months of Screening or currently has functioning implantable electric stimulator.
6. Nasogastric, percutaneous endoscopic gastrostomy, or percutaneous endoscopic jejunostomy feeding tube or inpatient hospitalization for gastroparesis within 2 weeks before the Screening Visit.
7. Required parenteral nutrition for treatment of gastroparesis within 2 months before the Screening Visit.
8. Previous diagnosis of gastric bezoar (the presence of retained liquid, bile, or small amounts of poorly organized food residue is permitted).
9. Poor control of diabetes within 30 days prior to randomization, including diabetic ketoacidosis, hypoglycemia requiring medical intervention, admission for control of diabetes or diabetic complications.
10. Elevated serum prolactin (>upper limit of normal [ULN]) at Screening.
11. Has concurrent hypogonadism, current clinically significant menstrual abnormalities, such as amenorrhea or oligomenorrhea, or other clinical features of hyperprolactinemia such as galactorrhea or gynecomastia.
12. Has acute or chronic liver disease meeting any of the criteria described below:

    * Has an alanine aminotransferase (ALT), aspartate aminotransferase (AST) or total bilirubin >2.0 times the ULN.
    * Has pre-existing liver cirrhosis that meets Child-Pugh Class B (moderate; total score 7 to 9 points) or C (severe; total score 10 to 15 points) (see Appendix B).
    * Has acute or chronic hepatitis B or C virus infection, manifesting as one of the following at screening:
    * Positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). NOTE: if a participants tests negative for HBsAg, but positive for HBcAb, the participant would be eligible if the Investigator has documentation of other test results showing that the participant does not have active hepatitis B infection.
    * Participants with positive hepatitis C antibody (HCV IgG) and quantitative HCV polymerase chain reaction (PCR). HCV PCR is performed only if HCV IgG is positive.
13. Has renal impairment, defined as a lower limit of (estimated glomerular filtration rate [eGFR]) <30 mL/min at screening visit.
14. Has active neoplastic disease or history of neoplastic disease within 5 years of screening visit (except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the uterine cervix that has been definitively treated with standard of care approaches).
15. Uncontrolled or poorly controlled medical or psychiatric comorbidities which might affect their ability to participate in the study.
16. Has known COVID-19 infection, or suspected COVID-19 infection (as assessed by the investigator).
17. Signs/symptoms or history of extrapyramidal system disease and other clinically relevant CNS or neuropsychiatric disease including but not limited to tardive dyskinesia, neuroleptic malignant syndrome, acute dystonia, parkinsonian like symptoms, severe mental depression, and history of suicide attempt.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2018-10-14 (Actual); Primary Completion 2021-06-14 (Actual); Study Completion 2021-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (108):
- United States (66):
  - Digestive Health Specialists of the Southeast, Dothan, Alabama
  - Del Sol Research Management, Tucson, Arizona
  - GW Research, Chula Vista, California
  - Trial Connections - New Hope Research Development, Corona, California
  - Paragon Rx Clinical - Garden Grove, Garden Grove, California
  - Torrance Clinical Research Institute Inc., Lomita, California
  - California Medical Research Associates, Northridge, California
  - ISS - Conquest Clinical Research, Orange, California
  - Precision Research Institute, San Diego, California
  - Connecticut Clinical Research Foundation, Bristol, Connecticut
  - ISS - Innovative Research of West Florida, Clearwater, Florida
  - Elias Research Associates - Direct Helpers Research Center - Hialeah, Hialeah, Florida
  - International Research Associates, Hialeah, Florida
  - Palmetto Research, Hialeah, Florida
  - Homestead Associates in Research, Homestead, Florida
  - Gastroenterology Associates - Crystal River, Inverness, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Baptist Diabetes Associates Research, Miami, Florida
  - PharmaSouth Research, Miami, Florida
  - Miami Dade Medical Research Institute, Miami, Florida
  - Anchor Medical Research, Miami, Florida
  - Advanced Research Institute - New Port Richey, New Port Richey, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Summit Clinical Research, Athens, Georgia
  - Digestive Healthcare of Georgia - Atlanta, Atlanta, Georgia
  - DM Clinical Research - Southwest Gastroenterology - Oak Lawn, Oak Lawn, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Tri-State Gastroenterology Associates, Crestview Hills, Kentucky
  - Gastro Center of Maryland, Columbia, Maryland
  - MGH Digestive Healthcare, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - West Roxbury, West Roxbury, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - Gastroenterology Associates of Western Michigan, Wyoming, Michigan
  - Gastrointestinal Associates and Endoscopy Center, Flowood, Mississippi
  - Montana Medical Research, Missoula, Montana
  - Lovelace Scientific Resources - Albuquerque, Albuquerque, New Mexico
  - NY Scientific, Brooklyn, New York
  - Long Island Gastrointestinal Research Group, Great Neck, New York
  - Atrium Health, Charlotte, North Carolina
  - Chevy Chase Clinical Research, Concord, North Carolina
  - Fayetteville Gastroenterology Associates, Fayetteville, North Carolina
  - Carolina Digestive Diseases, Greenville, North Carolina
  - Wake Research Associates, Raleigh, North Carolina
  - PMG Research of Salisbury, Salisbury, North Carolina
  - Trial Management Associates, Wilmington, North Carolina
  - Gastroenterology Associates of the Piedmont, Winston-Salem, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Providence Health Partners - Center for Clinical Research, Dayton, Ohio
  - Elite Research - Lynn Institute of Stillwater, Stillwater, Oklahoma
  - Options Health Research, Tulsa, Oklahoma
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Digestive Disease Associates - Wyomissin, Wyomissing, Pennsylvania
  - ClinSearch, Chattanooga, Tennessee
  - Clinical Research Solutions - Jackson, Jackson, Tennessee
  - New Phase Research and Development, Knoxville, Tennessee
  - Quality Medical Research, Nashville, Tennessee
  - Texas Tech University Health Sciences Center - El Paso, El Paso, Texas
  - Spring Gastroenterology Associates - Houston, Houston, Texas
  - Biopharma Informatic Houston 1, Houston, Texas
  - Biopharma Informatic Houston 2, Houston, Texas
  - Rio Grande Gastroenterology, McAllen, Texas
  - Clinical Associates in Research Therapeutics of America, San Antonio, Texas
  - Sun Research Institute, San Antonio, Texas
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
- Belgium (7):
  - Universiteit Antwerpen, Edegem, Antwerpen
  - Universitair Ziekenhuis Leuven, Leuven, Flemish Brabant
  - Algemeen Ziekenhuis Sint-Lucas, Bruges, West-vlaanderen
  - AZ Groeninge Campus Kennedylaan, Kortrijk, West-vlaanderen
  - Hopital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Universiteit Gent, Ghent
- Japan (29):
  - Tokai Memorial Hospital, Kasugai-shi, Aichi-ken
  - Meitetsu Hospital, Nagoya, Aichi-ken
  - Chubu-Rosai Hospital, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - Tokatsu Tsujinaka Hospital, Abiko, Chiba
  - Matsuyama Shimin Hospital, Matsuyama, Ehime
  - Hatakeyama Clinic, Fukuoka, Fukuoka
  - Oishi Clinic, Kasuya-gun, Fukuoka
  - Igarashi Internal Medicine Surgery Clinic, Kōriyama, Fukushima
  - Asahi University Hospital, Gifu, Gifu
  - Nakamura Digestive Organ Internal Medicine Clinic, Bibai, Hokkaido
  - Akakura GI Clinic, Sapporo, Hokkairdo
  - Hyogo Prefectural Nishinomiya Hospital, Nishinomiya, Hyōgo
  - Hyogo College of Medicine Hospital, Nishinomiya, Hyōgo
  - Takarazuka City Hospital, Takarazuka-shi, Hyōgo
  - Hitachi, Ltd. Hitachinaka General Hospital, Hitachi, Ibaraki
  - Minami Akatsuka Clinic, Mito, Ibaraki
  - Tsuchiura Beryl Clinic, Tsuchiura, Ibaraki
  - Medical Corporation Shintoukai Yokohama Minoru Clinic, Yokohama, Kanagawa
  - Takatsuki Red Cross Hospital, Takatsuki-shi, Osaka
  - Medical Corporation Kumagaya General Hospital, Kumagaya, Saitama
  - Wakasa Clinic, Tokorozawa, Saitama
  - Community Hospital Koga Hospital, Yaizu, Shizuoka
  - Shimokitazawa Tomo Clinic, Setagaya-Ku, Tokyo
  - Morinaga Ueno Clinic, Kumamoto
  - Ijinkai Takeda General Hospital, Kyoto
  - Okayama Saiseikai General Hospital, Okayama
  - Medical Corporation Kamata Clinic, Saitama
  - Gastroenterology and Internal Medicine, Oizumi Medical Clinic, Yamagata
- Poland (6):
  - VITAMED Galaj i Cichomski spolka jawna, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Centrum Medyczne Clw-Med Aneta Cichomska i Joanna uka-Wendrowska sp.j., Grudziądz, Kuyavian-Pomeranian Voivodeship
  - Bodyclinic, Warsaw, Masovian Voivodeship
  - Centrum Medyczne Lukamed Joanna Luka, Chojnice, Pomeranian Voivodeship
  - Endoskopia, Sopot
  - Niepubliczny Zaklad Opieki Zdrowotnej - Witamed Poradnia Diabetolo, Kielce, Świętokrzyskie Voivodeship

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Tack J, McCallum R, Kuo B, Huh SY, Zhang Y, Chen YJ, Mehrotra S, Parkman HP. Randomized clinical trial: A phase 2b controlled study of the efficacy and safety of trazpiroben (TAK-906) for idiopathic or diabetic gastroparesis. Neurogastroenterol Motil. 2023 Oct;35(10):e14652. doi: 10.1111/nmo.14652. Epub 2023 Aug 3. PMID 37533380
- [Derived] Yamaguchi T, Kudou K, Okamoto H, Chen C, Whiting R, Sekino H. Evaluating the Safety, Tolerability, and Disposition of Trazpiroben, a D2 /D3 Receptor Antagonist: Phase I Single- and Multiple-Ascending Dose Studies in Healthy Japanese Participants. Clin Pharmacol Drug Dev. 2022 Jun;11(6):695-706. doi: 10.1002/cpdd.1057. Epub 2021 Dec 29. PMID 34967147
- See also: Related Info — https://clinicaltrials.takeda.com/study-detail/5f6b60354db2bf003ab4a062

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with symptomatic idiopathic or diabetic gastroparesis took part in the study at 73 investigative sites in Belgium, Poland, Japan and the United States from 14 October 2018 to 15 July 2021.
Pre-assignment Details: Participants receive TAK-906 5 mg, 25 mg, 50 mg Maleate or placebo in 1:1:1:1 ratio until protocol amendment 8 was implemented. As pre-specified in protocol amendment 8 further randomization TAK-906 5 mg arm was discontinued and remaining enrolled participants were randomized into TAK-906 25 mg, TAK-906 50 mg Maleate or placebo in 1:1:1 ratio.
Period: Overall Study
Arm/Group | Placebo | TAK-906 Maleate 5 mg | TAK-906 Maleate 25 mg | TAK-906 Maleate 50 mg
Started | 73 | 23 | 72 | 74
Completed | 67 | 21 | 67 | 72
Not Completed | 6 | 2 | 5 | 2
Not completed — Adverse Event | 1 | 0 | 1 | 0
Not completed — Protocol Deviation | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 3 | 0 | 0 | 2
Not completed — Voluntary Withdrawal | 2 | 1 | 3 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Randomized Set included all participants who were randomized.
Groups:
- Placebo: TAK-906 maleate placebo-matching capsules, orally, BID for up to 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Placebo | TAK-906 Maleate 5 mg | TAK-906 Maleate 25 mg | TAK-906 Maleate 50 mg | Total
Number analyzed (Participants) | 73 | 23 | 72 | 74 | 242
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.1 (14.22) | 56.3 (14.32) | 56.4 (13.31) | 53.4 (15.09) | 55.7 (14.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 19 | 61 | 49 | 183
  Male | 19 | 4 | 11 | 25 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 14 | 38 | 28 | 110
  Not Hispanic or Latino | 42 | 9 | 34 | 45 | 130
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 8 | 4 | 12 | 15 | 39
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 10 | 1 | 4 | 11 | 26
  White | 54 | 18 | 55 | 45 | 172
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 3 | 0 | 3 | 3 | 9
  Japan | 8 | 4 | 10 | 13 | 35
  Poland | 2 | 0 | 2 | 2 | 6
  United States of America | 60 | 19 | 57 | 56 | 192
Height [Mean (Standard Deviation); unit: centimetres (cm)] | 164.17 (10.238) | 164.43 (9.178) | 161.32 (7.313) | 166.12 (8.841) | 163.94 (9.054)
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 79.35 (16.383) | 82.62 (17.021) | 71.97 (16.261) | 78.77 (15.201) | 77.29 (16.36)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI was calculated as weight (kg) divided by square of height (m^2).
  kg/m^2 | 29.35 (5.003) | 30.48 (5.606) | 27.61 (5.835) | 28.52 (4.934) | 28.69 (5.343)
Smoking Classification [Count of Participants; unit: Participants]
  Participant has Never Smoked | 51 | 18 | 57 | 54 | 180
  Participant is a Current Smoker | 10 | 1 | 7 | 5 | 23
  Participant is an Ex-smoker | 12 | 4 | 8 | 15 | 39
ANMS GCSI-DD Composite Score [Mean (Full Range); unit: score on a scale] — American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary(ANMS GCSI-DD):patient-reported outcome instrument for symptom-based clinical trial endpoint in gastroparesis. ANMS GCSI-DD composite score: nausea, early satiety, upper abdominal pain and postprandial fullness.Daily composite score was calculated by summing scores on 4 symptom items(nausea, early satiety, postprandial fullness, and upper abdominal pain)/4 (number of items within composite score). ANMS GCSI-DD daily composite score ranged from 0 to 4 with higher scores=greater symptom severity. Population: FAS included all participants who were randomized, received at least 1 dose of study drug, and have a baseline value and at least 1 valid postbaseline value for assessment of primary efficacy.
  score on a scale | 2.59 [2.0 to 4.0] | 2.77 [2.0 to 3.8] | 2.57 [2.0 to 4.0] | 2.64 [2.0 to 4.0] | 2.62 [2 to 4]
ANMS GCSI-DD Nausea Symptom Score [Mean (Full Range); unit: score on a scale] — ANMS GCSI-DD is a patient-reported outcome instrument for a symptom-based clinical trial endpoint in gastroparesis. The ANMS GCSI-DD assesses nausea, early satiety, postprandial fullness, and upper abdominal pain on a severity score calculated from a 5-point Likert scale. The ANMS GCSI-DD nausea symptom score ranged from 0 to 4 with higher scores reflecting greater symptom severity. Population: FAS included all participants who were randomized, received at least 1 dose of study drug, and have a baseline value and at least 1 valid postbaseline value for assessment of primary efficacy.
  score on a scale | 2.80 [1.6 to 4.0] | 2.85 [1.7 to 4.0] | 2.70 [1.6 to 4.0] | 2.72 [1.9 to 4.0] | 2.75 [1.6 to 4]
ANMS GCSI-DD Early Satiety Symptom Score [Mean (Full Range); unit: score on a scale] — ANMS GCSI-DD is a patient-reported outcome instrument for a symptom-based clinical trial endpoint in gastroparesis. The ANMS GCSI-DD assesses nausea, early satiety, postprandial fullness, and upper abdominal pain on a severity score calculated from a 5-point Likert scale. The ANMS GCSI-DD early satiety symptom score ranged from 0 to 4 with higher scores reflecting greater symptom severity. Population: FAS included all participants who were randomized, received at least 1 dose of study drug, and have a baseline value and at least 1 valid postbaseline value for assessment of primary efficacy.
  score on a scale | 2.80 [1.3 to 4.0] | 2.97 [2.0 to 4.0] | 2.82 [1.3 to 4.0] | 2.82 [1.9 to 4.0] | 2.83 [1.3 to 4.0]
ANMS GCSI-DD Postprandial Fullness Symptom Score [Mean (Full Range); unit: score on a scale] — ANMS GCSI-DD is a patient-reported outcome instrument for a symptom-based clinical trial endpoint in gastroparesis. The ANMS GCSI-DD assesses nausea, early satiety, postprandial fullness, and upper abdominal pain on a severity score calculated from a 5-point Likert scale. The ANMS GCSI-DD postprandial fullness symptom score ranged from 0 to 4 with higher scores reflecting greater symptom severity. Population: FAS included all participants who were randomized, received at least 1 dose of study drug, and have a baseline value and at least 1 valid postbaseline value for assessment of primary efficacy.
  score on a scale | 2.99 [2.0 to 4.0] | 3.16 [2.1 to 4.0] | 2.98 [2.0 to 4.0] | 3.08 [2.0 to 4.0] | 3.03 [2.0 to 4.0]
ANMS GCSI-DD Upper Abdominal Pain Symptom Score [Mean (Full Range); unit: score on a scale] — ANMS GCSI-DD is a patient-reported outcome instrument for a symptom-based clinical trial endpoint in gastroparesis. The ANMS GCSI-DD assesses nausea, early satiety, postprandial fullness, and upper abdominal pain on a severity score calculated from a 5-point Likert scale. The ANMS GCSI-DD upper abdominal pain symptom score ranged from 0 to 4 with higher scores reflecting greater symptom severity. Population: FAS included all participants who were randomized, received at least 1 dose of study drug, and have a baseline value and at least 1 valid postbaseline value for assessment of primary efficacy.
  score on a scale | 1.76 [0.0 to 4.0] | 2.11 [0.1 to 4.0] | 1.77 [0.0 to 4.0] | 1.94 [0.0 to 3.9] | 1.85 [0.0 to 4.0]
ANMS GCSI-DD Recorded Vomiting Frequency [Mean (Full Range); unit: vomiting episodes/day] — Vomiting frequency was collected as the number of times a participant vomited in a 24-hour period i.e., vomiting episodes using the ANMS GCSI-DD. The daily score was averaged over 7 days. Higher scores indicate more severe symptoms. Population: FAS included all participants who were randomized, received at least 1 dose of study drug, and have a baseline value and at least 1 valid postbaseline value for assessment of primary efficacy.
  vomiting episodes/day | 1.41 [0.0 to 11.4] | 0.73 [0.0 to 1.9] | 1.25 [0.0 to 7.9] | 1.18 [0.0 to 11.0] | 1.23 [0.0 to 11.4]
ANMS GCSI-DD Overall Severity of Gastroparesis Symptoms Score [Mean (Full Range); unit: score on a scale] — The overall severity of gastroparesis symptoms is the participant report of the overall severity rating of their symptoms as entered daily in the ANMS GCSI-DD and at time of visit. Severity was rated on a 0 (none) to 4 (very severe) scale. Higher score values indicated more severe symptoms. Population: FAS included all participants who were randomized, received at least 1 dose of study drug, and have a baseline value and at least 1 valid postbaseline value for assessment of primary efficacy.
  score on a scale | 2.90 [2.0 to 4.0] | 3.07 [2.0 to 4.0] | 2.86 [1.4 to 4.0] | 2.86 [1.4 to 4.0] | 2.89 [1.4 to 4.0]
Bloating Severity Scale Score [Mean (Full Range); unit: score on a scale] — The bloating severity scale was scored from 0 to 4 (where 0 = no symptom and 4 = severe symptom). The daily total score can range from 0 to 4 with higher scores reflecting greater symptom severity. Population: FAS included all participants who were randomized, received at least 1 dose of study drug, and have a baseline value and at least 1 valid postbaseline value for assessment of primary efficacy.
  score on a scale | 2.86 [2.0 to 4.0] | 3.13 [2.0 to 4.0] | 2.89 [1.1 to 4.0] | 2.91 [1.7 to 4.0] | 2.91 [1.1 to 4.0]
ANMS GCSI-DD Total Score [Mean (Full Range); unit: score on a scale] — Daily total score was calculated by summing scores on each of the 5 symptom items in ANMS GCSI-DD (nausea, early satiety, postprandial fullness, upper abdominal pain and vomiting) plus the bloating severity item and then dividing by 6. When calculating total score, vomiting frequency was scored from 0 to 4 (where 0=no vomiting and 4=four or more episodes of vomiting). The daily total score can range from 0 to 4 with higher scores reflecting greater symptom severity. Population: FAS included all participants who were randomized, received at least 1 dose of study drug, and have a baseline value and at least 1 valid postbaseline value for assessment of primary efficacy.
  score on a scale | 2.40 [1.7 to 3.6] | 2.49 [1.7 to 3.4] | 2.37 [1.5 to 4.0] | 2.41 [1.7 to 3.8] | 2.40 [1.5 to 4.0]
PAGI-SYM Total Score [Mean (Full Range); unit: score on a scale] — The patient assessment of upper gastrointestinal disorders-symptom severity index (PAGI-SYM) total score is defined as the mean of 6 PAGI-SYM subscale scores from 20 items. A 6-point Likert response scale, ranging from 0 (none) to 5 (very severe), is used to measure symptom severity in patients with upper GI disorders. Population: FAS included all participants who were randomized, received at least 1 dose of study drug, and have a baseline value and at least 1 valid postbaseline value for assessment of primary efficacy.
  score on a scale | 3.13 [0.1 to 4.9] | 3.33 [2.1 to 4.7] | 3.05 [1.7 to 4.7] | 3.13 [1.0 to 4.9] | 3.13 [0.1 to 4.9]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the American Neurogastroenterology and Motility Society Gastroparesis Cardinal Symptom Index-Daily Diary (ANMS GCSI-DD) Composite Score at Week 12 of the Treatment Period
Description: ANMS GCSI-DD is a patient-reported outcome instrument for a symptom-based clinical trial endpoint in gastroparesis. The ANMS GCSI-DD composite score included score of nausea, early satiety, upper abdominal pain, and postprandial fullness. The severity scores of these symptoms range from 0 (none) to 4 (very severe). The daily composite score was calculated by summing the scores on the 4 symptom items (nausea, early satiety, postprandial fullness, and upper abdominal pain) and then dividing by 4, that is the number of items within the composite score. Thus, the maximum daily composite score was (4 symptoms × maximum score 4 divided by 4) = 16/4 = 4. The ANMS GCSI-DD daily composite score ranged from 0 to 4 with higher scores reflecting greater symptom severity. The negative change from baseline indicates improvement. Mixed-effects Model for Repeated Measures (MMRM) was used for the analysis.
Time Frame: Baseline and Week 12
Population: FAS included all participants who were randomized, received at least 1 dose of study drug, and have a baseline value and at least 1 valid postbaseline value for assessment of primary efficacy.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-906 Maleate 5 mg | TAK-906 Maleate 25 mg | TAK-906 Maleate 50 mg
Number analyzed (Participants) | 73 | 23 | 72 | 74
score on a scale | -1.19 (0.120) | -1.11 (0.219) | -1.17 (0.120) | -1.21 (0.116)
Statistical Analysis 1: Comparison: Placebo vs TAK-906 Maleate 5 mg; Test type: Superiority; p = 0.618, MMRM — 1-sided p-values were obtained using MMRM Model. It was based on the one-sided alternative hypothesis testing that the treatment difference (TAK-906 - Placebo) in ANMS GCSI-DD composite score was <0; Least Square Mean Difference = 0.08, 90% CI 2-sided [-0.34 to 0.49], Standard Error of Mean 0.250 — MMRM included week, treatment, participant disease population (DG/IG), treatment-by-week interaction as fixed effects, baseline and baseline score-by-week interaction as covariates, with an unstructured working covariance matrix as default
Statistical Analysis 2: Comparison: Placebo vs TAK-906 Maleate 25 mg; Test type: Superiority; p = 0.533, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Square Mean Difference = 0.01, 90% CI 2-sided [-0.27 to 0.29], Standard Error of Mean 0.170 — MMRM model included week, treatment, participant disease population (DG/IG), treatment-by-week interaction as fixed effects, baseline and baseline score-by-week interaction as covariates, with an unstructured working covariance matrix as default
Statistical Analysis 3: Comparison: Placebo vs TAK-906 Maleate 50 mg; Test type: Superiority; p = 0.447, MMRM — [p-value comment as in outcome 1, analysis 1]; Least Square Mean Difference = -0.02, 90% CI 2-sided [-0.30 to 0.25], Standard Error of Mean 0.167 — [estimate comment as in outcome 1, analysis 2]

2. Secondary Outcome: Percentage of Participants With at Least 50% Reduction From Baseline in ANMS GCSI-DD Composite Score at Week 12
Description: ANMS GCSI-DD is a patient-reported outcome instrument for a symptom-based clinical trial endpoint in gastroparesis . The ANMS GCSI-DD composite score included score of nausea, early satiety, upper abdominal pain and postprandial fullness. The severity scores of these symptoms range from 0 (none) to 4 (very severe). The daily composite score was calculated by summing the scores on the 4 symptom items (nausea, early satiety, postprandial fullness, and upper abdominal pain) and then dividing by 4, that is the number of items within the composite score. Thus, the maximum daily composite score was (4 symptoms × maximum score 4 divided by 4) = 16/4 = 4. The ANMS GCSI-DD daily composite score ranged from 0 to 4 with higher scores reflecting greater symptom severity.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | TAK-906 Maleate 5 mg | TAK-906 Maleate 25 mg | TAK-906 Maleate 50 mg
Number analyzed (Participants) | 73 | 23 | 72 | 74
percentage of participants | 42.5 | 39.1 | 47.2 | 41.9
Statistical Analysis 1: Comparison: Placebo vs TAK-906 Maleate 5 mg; Test type: Superiority; p = 0.607, Logistic Regression; Odds Ratio (OR) = 0.87, 90% CI 2-sided [0.39 to 1.96] — Comparisons of TAK-906 to Placebo was based on logistic regression with at least 50% reduction of participants from baseline in weekly composite score with baseline composite score, disease population at randomization, and treatment as covariates
Statistical Analysis 2: Comparison: Placebo vs TAK-906 Maleate 25 mg; Test type: Superiority; p = 0.283, Logistic Regression; Odds Ratio (OR) = 1.21, 90% CI 2-sided [0.70 to 2.10] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs TAK-906 Maleate 50 mg; Test type: Superiority; p = 0.527, Logistic Regression; Odds Ratio (OR) = 0.98, 90% CI 2-sided [0.56 to 1.69] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Change From Baseline in the ANMS GCSI-DD Nausea Symptom Score at Week 12 of the Treatment Period
Description: ANMS GCSI-DD is a patient-reported outcome instrument for a symptom-based clinical trial endpoint in gastroparesis. The ANMS GCSI-DD assesses nausea, early satiety, postprandial fullness, and upper abdominal pain on a severity score calculated from a 5-point Likert scale. The ANMS GCSI-DD nausea symptom score ranged from 0 to 4 with higher scores reflecting greater symptom severity. The negative change from baseline indicates improvement. MMRM was used for analysis.
Time Frame: Baseline and Week 12
Population: FAS included all participants who were randomized, received at least 1 dose of study drug, and have a baseline value and at least 1 valid postbaseline value for assessment of primary efficacy. Overall number analyzed is the number of participants with data available for analysis.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-906 Maleate 5 mg | TAK-906 Maleate 25 mg | TAK-906 Maleate 50 mg
Number analyzed (Participants) | 50 | 15 | 55 | 58
score on a scale | -1.42 (0.134) | -1.36 (0.245) | -1.36 (0.133) | -1.40 (0.129)
Statistical Analysis 1: Comparison: Placebo vs TAK-906 Maleate 5 mg; Test type: Superiority; p = 0.584, MMRM — 1-sided p-values were obtained using MMRM Model. It was based on the one-sided alternative hypothesis testing that the treatment difference (TAK-906 - Placebo) in ANMS GCSI-DD nausea symptom score was <0; Least-Squares Mean Difference = 0.06, 90% CI 2-sided [-0.40 to 0.52], Standard Error of Mean 0.279 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs TAK-906 Maleate 25 mg; Test type: Superiority; p = 0.625, MMRM — [p-value comment as in outcome 3, analysis 1]; Least-Squares Mean Difference = 0.06, 90% CI 2-sided [-0.25 to 0.37], Standard Error of Mean 0.189 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs TAK-906 Maleate 50 mg; Test type: Superiority; p = 0.540, MMRM — [p-value comment as in outcome 3, analysis 1]; Least-Squares Mean Difference = 0.02, 90% CI 2-sided [-0.29 to 0.33], Standard Error of Mean 0.187 — [estimate comment as in outcome 1, analysis 2]

4. Secondary Outcome: Change From Baseline in the ANMS GCSI-DD Early Satiety Symptom Score at Week 12 of the Treatment Period
Description: ANMS GCSI-DD is a patient-reported outcome instrument for a symptom-based clinical trial endpoint in gastroparesis. The ANMS GCSI-DD assesses nausea, early satiety, postprandial fullness, and upper abdominal pain on a severity score calculated from a 5-point Likert scale. The ANMS GCSI-DD early satiety symptom score ranged from 0 to 4 with higher scores reflecting greater symptom severity. The negative change from Baseline indicated improvement. MMRM was used for the analysis.
Time Frame: Baseline and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-906 Maleate 5 mg | TAK-906 Maleate 25 mg | TAK-906 Maleate 50 mg
Number analyzed (Participants) | 50 | 15 | 55 | 58
score on a scale | -1.26 (0.136) | -1.25 (0.248) | -1.17 (0.135) | -1.33 (0.131)
Statistical Analysis 1: Comparison: Placebo vs TAK-906 Maleate 5 mg; Test type: Superiority; p = 0.510, MMRM — 1-sided p-values were obtained using MMRM Model. It was based on the one-sided alternative hypothesis testing that the treatment difference (TAK-906 - Placebo) in ANMS GCSI-DD early satiety symptom score was <0; Least-Squares Mean Difference = 0.01, 90% CI 2-sided [-0.46 to 0.47], Standard Error of Mean 0.283 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs TAK-906 Maleate 25 mg; Test type: Superiority; p = 0.674, MMRM — [p-value comment as in outcome 4, analysis 1]; Least-Squares Mean Difference = 0.09, 90% CI 2-sided [-0.23 to 0.40], Standard Error of Mean 0.192 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs TAK-906 Maleate 50 mg; Test type: Superiority; p = 0.367, MMRM — [p-value comment as in outcome 4, analysis 1]; Least-Squares Mean Difference = -0.06, 90% CI 2-sided [-0.38 to 0.25], Standard Error of Mean 0.189 — [estimate comment as in outcome 1, analysis 2]

5. Secondary Outcome: Change From Baseline in the ANMS GCSI-DD Postprandial Fullness Symptom Score at Week 12 of the Treatment Period
Description: ANMS GCSI-DD is a patient-reported outcome instrument for a symptom-based clinical trial endpoint in gastroparesis. The ANMS GCSI-DD assesses nausea, early satiety, postprandial fullness, and upper abdominal pain on a severity score calculated from a 5-point Likert scale. The ANMS GCSI-DD postprandial fullness symptom score ranged from 0 to 4 with higher scores reflecting greater symptom severity. The negative change from baseline indicates improvement. MMRM was used for the analysis.
Time Frame: Baseline and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-906 Maleate 5 mg | TAK-906 Maleate 25 mg | TAK-906 Maleate 50 mg
Number analyzed (Participants) | 50 | 15 | 55 | 58
score on a scale | -1.32 (0.139) | -1.26 (0.253) | -1.27 (0.138) | -1.35 (0.134)
Statistical Analysis 1: Comparison: Placebo vs TAK-906 Maleate 5 mg; Test type: Superiority; p = 0.587, MMRM — 1-sided p-values were obtained using MMRM Model. It was based on the one-sided alternative hypothesis testing that the treatment difference (TAK-906 - Placebo) in ANMS GCSI-DD postprandial fullness symptom score was <0; Least-Squares Mean Difference = 0.06, 90% CI 2-sided [-0.41 to 0.54], Standard Error of Mean 0.289 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs TAK-906 Maleate 25 mg; Test type: Superiority; p = 0.600, MMRM — [p-value comment as in outcome 5, analysis 1]; Least-Squares Mean Difference = 0.05, 90% CI 2-sided [-0.27 to 0.37], Standard Error of Mean 0.196 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs TAK-906 Maleate 50 mg; Test type: Superiority; p = 0.446, MMRM — [p-value comment as in outcome 5, analysis 1]; Least-Squares Mean Difference = -0.03, 90% CI 2-sided [-0.34 to 0.29], Standard Error of Mean 0.193 — [estimate comment as in outcome 1, analysis 2]

6. Secondary Outcome: Change From Baseline in the ANMS GCSI-DD Upper Abdominal Pain Symptom Score at Week 12 of the Treatment Period
Description: ANMS GCSI-DD is a patient-reported outcome instrument for a symptom-based clinical trial endpoint in gastroparesis. The ANMS GCSI-DD assesses nausea, early satiety, postprandial fullness, and upper abdominal pain on a severity score calculated from a 5-point Likert scale. The ANMS GCSI-DD upper abdominal pain symptom score ranged from 0 to 4 with higher scores reflecting greater symptom severity. The negative change from baseline indicates improvement. MMRM was used for the analysis.
Time Frame: Baseline and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-906 Maleate 5 mg | TAK-906 Maleate 25 mg | TAK-906 Maleate 50 mg
Number analyzed (Participants) | 50 | 15 | 55 | 58
score on a scale | -0.72 (0.118) | -0.68 (0.214) | -0.90 (0.117) | -0.76 (0.114)
Statistical Analysis 1: Comparison: Placebo vs TAK-906 Maleate 5 mg; Test type: Superiority; p = 0.562, MMRM — 1-sided p-values were obtained using MMRM Model. It was based on the one-sided alternative hypothesis testing that the treatment difference (TAK-906 - Placebo) in ANMS GCSI-DD upper abdominal pain symptom score was <0; Least-Squares Mean Difference = 0.04, 90% CI 2-sided [-0.37 to 0.44], Standard Error of Mean 0.245 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs TAK-906 Maleate 25 mg; Test type: Superiority; p = 0.138, MMRM — [p-value comment as in outcome 6, analysis 1]; Least-Squares Mean Difference = -0.18, 90% CI 2-sided [-0.46 to 0.09], Standard Error of Mean 0.166 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs TAK-906 Maleate 50 mg; Test type: Superiority; p = 0.394, MMRM — [p-value comment as in outcome 6, analysis 1]; Least-Squares Mean Difference = -0.04, 90% CI 2-sided [-0.32 to 0.23], Standard Error of Mean 0.164 — [estimate comment as in outcome 1, analysis 2]

7. Secondary Outcome: Change From Baseline in the ANMS GCSI-DD Recorded Vomiting Frequency at Week 12 of the Treatment Period
Description: Vomiting frequency was collected as the number of times a participant vomited in a 24-hour period i.e., vomiting episodes using the ANMS GCSI-DD. The daily score was averaged over 7 days. Higher scores indicate more severe symptoms. MMRM was used for the analysis.
Time Frame: Baseline and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: vomiting episodes/day
Arm/Group | Placebo | TAK-906 Maleate 5 mg | TAK-906 Maleate 25 mg | TAK-906 Maleate 50 mg
Number analyzed (Participants) | 50 | 15 | 55 | 57
vomiting episodes/day | -0.71 (0.236) | -0.44 (0.421) | -0.48 (0.234) | -0.63 (0.231)
Statistical Analysis 1: Comparison: Placebo vs TAK-906 Maleate 5 mg; Test type: Superiority; p = 0.709, MMRM — 1-sided p-values were obtained using MMRM Model. It was based on the one-sided alternative hypothesis testing that the treatment difference (TAK-906 - Placebo) in ANMS GCSI-DD recorded vomiting frequency was <0; Least-Squares Mean Difference = 0.27, 90% CI 2-sided [-0.53 to 1.07], Standard Error of Mean 0.484 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs TAK-906 Maleate 25 mg; Test type: Superiority; p = 0.760, MMRM — [p-value comment as in outcome 7, analysis 1]; Least-Squares Mean Difference = 0.24, 90% CI 2-sided [-0.31 to 0.78], Standard Error of Mean 0.332 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs TAK-906 Maleate 50 mg; Test type: Superiority; p = 0.591, MMRM — [p-value comment as in outcome 7, analysis 1]; Least-Squares Mean Difference = 0.08, 90% CI 2-sided [-0.47 to 0.62], Standard Error of Mean 0.330 — [estimate comment as in outcome 1, analysis 2]

8. Secondary Outcome: Change From Baseline in the ANMS GCSI-DD Overall Severity of Gastroparesis Symptoms Score at Week 12 of the Treatment Period
Description: The overall severity of gastroparesis symptoms is the participant report of the overall severity rating of their symptoms as entered daily in the ANMS GCSI-DD and at time of visit. Severity was rated on a 0 (none) to 4 (very severe) scale. Higher score values indicated more severe symptoms. MMRM was used for the analysis.
Time Frame: Baseline and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-906 Maleate 5 mg | TAK-906 Maleate 25 mg | TAK-906 Maleate 50 mg
Number analyzed (Participants) | 50 | 15 | 55 | 58
score on a scale | -1.20 (0.130) | -1.02 (0.237) | -1.22 (0.129) | -1.25 (0.125)
Statistical Analysis 1: Comparison: Placebo vs TAK-906 Maleate 5 mg; Test type: Superiority; p = 0.742, MMRM — 1-sided p-values were obtained using MMRM Model. It was based on the one-sided alternative hypothesis testing that the treatment difference (TAK-906 - Placebo) in ANMS GCSI-DD overall severity of gastroparesis symptoms score was <0; Least-Squares Mean Difference = 0.18, 90% CI 2-sided [-0.27 to 0.62], Standard Error of Mean 0.270 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs TAK-906 Maleate 25 mg; Test type: Superiority; p = 0.461, MMRM — [p-value comment as in outcome 8, analysis 1]; Least-Squares Mean Difference = -0.02, 90% CI 2-sided [-0.32 to 0.28], Standard Error of Mean 0.183 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs TAK-906 Maleate 50 mg; Test type: Superiority; p = 0.376, MMRM — [p-value comment as in outcome 8, analysis 1]; Least-Squares Mean Difference = -0.06, 90% CI 2-sided [-0.36 to 0.24], Standard Error of Mean 0.181 — [estimate comment as in outcome 1, analysis 2]

9. Secondary Outcome: Change From Baseline in the ANMS GCI-DD Bloating Severity Scale Score at Week 12 of the Treatment Period
Description: The bloating severity scale was scored from 0 to 4 (where 0 = no symptom and 4 = severe symptom). The daily total score can range from 0 to 4 with higher scores reflecting greater symptom severity. The negative change from baseline indicates improvement. MMRM was used for analysis.
Time Frame: Baseline and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-906 Maleate 5 mg | TAK-906 Maleate 25 mg | TAK-906 Maleate 50 mg
Number analyzed (Participants) | 50 | 15 | 55 | 58
score on a scale | -1.15 (0.137) | -1.09 (0.250) | -1.26 (0.136) | -1.16 (0.132)
Statistical Analysis 1: Comparison: Placebo vs TAK-906 Maleate 5 mg; Test type: Superiority; p = 0.591, MMRM — 1-sided p-values were obtained using MMRM Model. It was based on the one-sided alternative hypothesis testing that the treatment difference (TAK-906 - Placebo) in ANMS GCSI-DD bloating severity scale score was <0; Least-Squares Mean Difference = 0.07, 90% CI 2-sided [-0.41 to 0.54], Standard Error of Mean 0.286 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs TAK-906 Maleate 25 mg; Test type: Superiority; p = 0.291, MMRM — [p-value comment as in outcome 9, analysis 1]; Least-Squares mean Difference = -0.11, 90% CI 2-sided [-0.43 to 0.21], Standard Error of Mean 0.193 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs TAK-906 Maleate 50 mg; Test type: Superiority; p = 0.476, MMRM — [p-value comment as in outcome 9, analysis 1]; Least-Squares Mean Difference = -0.01, 90% CI 2-sided [-0.33 to 0.30], Standard Error of Mean 0.191 — [estimate comment as in outcome 1, analysis 2]

10. Secondary Outcome: Change From Baseline in the ANMS GCSI-DD Total Score at Week 12 of the Treatment Period
Description: Daily total score was calculated by summing scores on each of the 5 symptom items in ANMS GCSI-DD (nausea, early satiety, postprandial fullness, upper abdominal pain and vomiting) plus the bloating severity item and then dividing by 6. When calculating total score, vomiting frequency was scored from 0 to 4 (where 0=no vomiting and 4=four or more episodes of vomiting). The daily total score can range from 0 to 4 with higher scores reflecting greater symptom severity. MMRM was used for analyses.
Time Frame: Baseline and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-906 Maleate 5 mg | TAK-906 Maleate 25 mg | TAK-906 Maleate 50 mg
Number analyzed (Participants) | 50 | 15 | 55 | 58
score on a scale | -1.10 (0.108) | -1.00 (0.196) | -1.09 (0.107) | -1.11 (0.104)
Statistical Analysis 1: Comparison: Placebo vs TAK-906 Maleate 5 mg; Test type: Superiority; p = 0.675, MMRM — 1-sided p-values were obtained using MMRM Model. It was based on the one-sided alternative hypothesis testing that the treatment difference (TAK-906 - Placebo) in ANMS GCSI-DD total score was <0; Least-Squares Mean Difference = 0.10, 90% CI 2-sided [-0.27 to 0.47], Standard Error of Mean 0.224 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs TAK-906 Maleate 25 mg; Test type: Superiority; p = 0.531, MMRM — [p-value comment as in outcome 10, analysis 1]; Least-Squares Mean Difference = 0.01, 90% CI 2-sided [-0.24 to 0.26], Standard Error of Mean 0.152 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Placebo vs TAK-906 Maleate 50 mg; Test type: Superiority; p = 0.473, MMRM — [p-value comment as in outcome 10, analysis 1]; Least-Squares Mean Difference = -0.01, 90% CI 2-sided [-0.26 to 0.24], Standard Error of Mean 0.150 — [estimate comment as in outcome 1, analysis 2]

11. Secondary Outcome: Percentage of Symptomatic Weeks
Description: Symptomatic weeks are weeks with average composite symptom score assessed as >mild [ANMS GCSI-DD score ≥2] during 12 weeks of treatment. Analysis of variance (ANOVA) was used for the analysis.
Time Frame: Up to 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: percentage of weeks
Arm/Group | Placebo | TAK-906 Maleate 5 mg | TAK-906 Maleate 25 mg | TAK-906 Maleate 50 mg
Number analyzed (Participants) | 73 | 23 | 72 | 74
percentage of weeks | 54.89 (4.746) | 46.42 (8.474) | 50.03 (4.781) | 51.31 (4.714)
Statistical Analysis 1: Comparison: Placebo vs TAK-906 Maleate 5 mg; Test type: Superiority; p = 0.192, ANOVA — The 1-sided p-value was based on the one-sided alternative hypothesis testing that the treatment difference (TAK-906 -Placebo) in symptomatic weeks was <0; Least-Squares Mean Difference = -8.47, 90% CI 2-sided [-24.50 to 7.57], Standard Error of Mean 9.710
Statistical Analysis 2: Comparison: Placebo vs TAK-906 Maleate 25 mg; Test type: Superiority; p = 0.236, ANOVA — The 1-sided p-value was based on the one-sided alternative hypothesis testing that the treatment difference (TAK-906 - Placebo) in symptomatic weeks was <0; Least-Squares Mean Difference = -4.85, 90% CI 2-sided [-15.98 to 6.27], Standard Error of Mean 6.736
Statistical Analysis 3: Comparison: Placebo vs TAK-906 Maleate 50 mg; Test type: Superiority; p = 0.297, ANOVA — [p-value comment as in outcome 11, analysis 2]; Least-Squares Mean Difference = -3.58, 90% CI 2-sided [-14.62 to 7.47], Standard Error of Mean 6.689

12. Secondary Outcome: Change From Baseline in the Patient Assessment of Upper Gastrointestinal Disorders-Symptom Severity Index (PAGI-SYM) Total Score at Week 12 of the Treatment Period
Description: The PAGI-SYM total score is defined as the mean of 6 PAGI-SYM subscale scores from 20 items. A 6-point Likert response scale, ranging from 0 (none) to 5 (very severe), is used to measure symptom severity in participants with upper GI disorders. The negative change from baseline indicates improvement. MMRM was used for analysis.
Time Frame: Baseline and Week 12
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-906 Maleate 5 mg | TAK-906 Maleate 25 mg | TAK-906 Maleate 50 mg
Number analyzed (Participants) | 57 | 16 | 54 | 60
score on a scale | -1.33 (0.141) | -1.25 (0.265) | -1.51 (0.142) | -1.57 (0.136)
Statistical Analysis 1: Comparison: Placebo vs TAK-906 Maleate 5 mg; Test type: Superiority; p = 0.601, MMRM — 1-sided p-values were obtained using MMRM of PAGI-SYM total score. It was based on the one-sided alternative hypothesis testing that the treatment difference (TAK-906 - Placebo) in PAGI-SYM total score was <0; Least-Squares Mean Difference = 0.08, 90% CI 2-sided [-0.42 to 0.57], Standard Error of Mean 0.300 — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Placebo vs TAK-906 Maleate 25 mg; Test type: Superiority; p = 0.181, MMRM — [p-value comment as in outcome 12, analysis 1]; Least-Squares Mean Difference = -0.18, 90% CI 2-sided [-0.51 to 0.15], Standard Error of Mean 0.200 — MMRM model includes week, treatment, participant disease population (DG/IG), treatment-by-week interaction as fixed effects, baseline and baseline score-by-week interaction as covariates, with an unstructured working covariance matrix as default
Statistical Analysis 3: Comparison: Placebo vs TAK-906 Maleate 50 mg; Test type: Superiority; p = 0.114, MMRM — [p-value comment as in outcome 12, analysis 1]; Least-Squares Mean Diferrence = -0.24, 90% CI 2-sided [-0.56 to 0.09], Standard Error of Mean 0.196 — [estimate comment as in outcome 12, analysis 2]

ADVERSE EVENTS:
Time Frame: From the study start up to 30 days after end of treatment (up to approximately 16 weeks)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Safety data was collected for all participants evaluable for response.
Groups:
- TAK-906 5 mg: TAK-906 maleate 5 mg, capsules, orally, BID for up to 12 weeks.
- TAK-906 25 mg: TAK-906 maleate 25 mg, capsules, orally, BID for up to 12 weeks.
- TAK-906 50 mg: TAK-906 maleate 50 mg, capsules, orally, BID for up to 12 weeks.
Arm/Group | Placebo | TAK-906 5 mg | TAK-906 25 mg | TAK-906 50 mg
All-Cause Mortality (participants affected / at risk) | 0/73 | 0/23 | 0/72 | 0/74
Serious Adverse Events (participants affected / at risk) | 2/73 | 0/23 | 2/72 | 2/74
Other Adverse Events (participants affected / at risk) | 0/73 | 2/23 | 4/72 | 4/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=73) | TAK-906 5 mg (N=23) | TAK-906 25 mg (N=72) | TAK-906 50 mg (N=74)
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Intermittent claudication (Vascular disorders) | 0 | 0 | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=73) | TAK-906 5 mg (N=23) | TAK-906 25 mg (N=72) | TAK-906 50 mg (N=74)
Headache (Nervous system disorders) | 0 | 0 | 4 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 4
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2020-07-13): https://cdn.clinicaltrials.gov/large-docs/29/NCT03544229/Prot_000.pdf
  • Statistical Analysis Plan (2021-08-02): https://cdn.clinicaltrials.gov/large-docs/29/NCT03544229/SAP_001.pdf